# **Tanglewood Trail Walking Program in Rural Kentucky 2017**

| Institution/Site: | University of Kentucky |
|----------------------------------|------------------------|
| Document (Approval/Update) Date: | 05/16/17 |
| NCT Number: | NCT03495648 |
| IRB Number | 17-0283-P2H (43453) |
| Coversheet created: | 8/2/21 |

| For ORI Use Only: |
|-------------------|

Consent to Participate in a Research Study

# **Tanglewood Trail Walking Program**

#### WHY ARE YOU BEING INVITED TO TAKE PART IN THIS RESEARCH?

You are being invited to take part in a research study about how physical activity and fruit and vegetable consumption impact health. You are being invited to take part in this research study because you expressed interest, are at least 18 years of age, nonpregnant and in the event that you are randomized into the walking group you are in good enough health to walk 1 mile the majority of Saturday mornings June thru August 2017. If you volunteer to take part in this study, you will be one of about 100 people to do so.

#### WHO IS DOING THE STUDY?

The person in charge of this study is Dawn Brewer, PhD, RDN, LD of University of Kentucky, Department of Dietetics and Human Nutrition. There may be other people on the research team assisting at different times during the study.

#### WHAT IS THE PURPOSE OF THIS STUDY?

By doing this study, we hope to learn if adults who regularly attend a walking group and/or the farmer's market experience increases in physical activity, fruit and vegetable intake, community engagement, and biomarkers associated with adulthood chronic disease.

# ARE THERE REASONS WHY YOU SHOULD NOT TAKE PART IN THIS STUDY?

If you are under 18 years old, pregnant or unable to walk 1 mile the majority of Saturday mornings, you should not participate in this study. While we understand that you may not be able to attend every Saturday morning walking group or the farmers market, but we encourage you to do your best to make it possible to be present each Saturday morning June thru August 2017.

# WHERE IS THE STUDY GOING TO TAKE PLACE AND HOW LONG WILL IT LAST?

The research procedures will be conducted at the parking lot near the community swimming pool in Whitesburg, Kentucky. You will be placed by chance into a walking group or a farmer's market group. If you are placed in the walking group, you will need to come to this parking lot near the community swimming pool 15 times during the study. If you are placed into the farmer's market group, you will need to come to this parking lot near the community swimming pool 2 times during the study for approximately 1 hour each time, and you will need to come to the Letcher County Farmer's Market 13 times (the amount of time you spend there is up to you). Each of those visits will take approximately 15 minutes (13 of the days) or up to one hour (2 of the days). You will walk to the Letcher County Farmer's Market 13 times (after meeting in the parking lot) and the amount of time you spend at the market is up to you. Regardless of which group you are in, you will also be asked to fill out a short, third survey in November 2017. This

survey should take you no longer than 10 minutes. The total amount of time you will be asked to volunteer for this study is no more than 15 hours over the next 4 months.

#### WHAT WILL YOU BE ASKED TO DO?

All participants will fill out a survey and have their weight, height, waist circumference, blood pressure, carotenoid status and finger stick cholesterol and A1c taken twice – once in May 2017, the second time in September 2017. You will be asked to fill out a shorter version of the survey in November 2017. Half of participants will be asked to report every Saturday morning to the parking lot near the community swimming pool to sign in and receive a voucher for the farmer's market. The other half of participants will report directly to the farmer's market to receive their voucher. All participants will turn in their voucher to the market manager, who will rip off the small end in return for \$10 worth of tokens to spend on fruits and vegetables at the farmer's market. The part of the voucher returned to you will ask you to do two things. First, you will be asked what fruits and vegetables, by color, you ate over the past week. Second, you will be asked to write down what fruits and vegetables you bought at the market that day. This voucher must be turned in to the market manager as you leave the market in order for you to receive your voucher the following week.

If you are placed into the farmer's market group, you can walk or drive to the market from any location you would like.

#### WHAT ARE THE POSSIBLE RISKS AND DISCOMFORTS?

To the best of our knowledge, the things you will be doing have no more risk of harm than you would experience in everyday life. The risks associated with finger stick readings are minimal and short term, but may include initial pain and tenderness. No participant will be stuck more than three times and all participants will receive band aids and proper attention and care. There are no risks associated with the use of a carotenoid scanner. Additionally, there is always the risk for unforeseeable risks.

#### WILL YOU BENEFIT FROM TAKING PART IN THIS STUDY?

There is no guarantee that you will get any benefit from taking part in this study. However, some people have experienced improved self-perceived health, a decrease in blood pressure, waist circumference, cholesterol, and a1c. Your willingness to take part, however, may, in the future, help society as a whole better understand this research topic.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any benefits or rights you would normally have if you choose not to volunteer. You can stop at any time during the study and still keep the benefits and rights you had before volunteering.

# IF YOU DON'T WANT TO TAKE PART IN THE STUDY, ARE THERE OTHER CHOICES?

If you do not want to be in the study, there are no other choices except not to take part in the study.

#### WHAT WILL IT COST YOU TO PARTICIPATE?

There are no costs associated with taking part in the study.

# WHO WILL SEE THE INFORMATION THAT YOU GIVE?

We will make every effort to keep confidential all research records that identify you to the extent allowed by law.

Your information will be combined with information from other people taking part in the study. When we write about the study to share it with other researchers, we will write about the combined information we have gathered. You will not be personally identified in these written materials. We may publish the results of this study; however, we will keep your name and other identifying information private.

We will make every effort to prevent anyone who is not on the research team from knowing that you gave us information, or what that information is. The collated data will only reveal summarized data without identifiable information. The de-identified data will be available electronically and stored on a password protected computer. The electronic document containing names with respective survey codes will be deleted after post-survey data has been collected and therefore will not be stored. The list will be deleted by January 2019. Any study materials and raw data will be retained for 6 years after study closure in a locked drawer within a locked office or on a password protected computer. The primary investigator and program manager assigned to the project and involved in data collection will have access to these items. Officials from the University of Kentucky or the National Institute of Health may look at or copy pertinent portions of records that identify you.

#### CAN YOUR TAKING PART IN THE STUDY END EARLY?

If you decide to take part in the study you still have the right to decide at any time that you no longer want to continue. You will not be treated differently if you decide to stop taking part in the study.

The individuals conducting the study may need to withdraw you from the study. This may occur if you are not able to follow the directions they give you, if they find that your being in the study is more risk than benefit to you, or if the agency funding the study decides to stop the study early for a variety of scientific reasons. You will be asked to have your height, weight, waist circumference, blood pressure, carotenoid status and finger stick cholesterol and A1c measured.

#### WHAT HAPPENS IF YOU GET HURT OR SICK DURING THE STUDY?

If you believe you are hurt or if you get sick because of something that is due to the study, you should call Dawn Brewer at 859-257-1661 immediately.

Dawn Brewer will determine what type of treatment, if any, that is best for you at that time.

It is important for you to understand that the University of Kentucky does not have funds set aside to pay for the cost of any care or treatment that might be necessary because you get hurt or sick while taking part in this study. Also, the University of Kentucky will not pay for any wages you may lose if you are harmed by this study.

You do not give up your legal rights by signing this form.

## WILL YOU RECEIVE ANY REWARDS FOR TAKING PART IN THIS STUDY?

All participants will receive a farmer's market t-shirt for their participation in May, a \$10 gift card for their participation in September, and \$10 farmers market voucher for every Saturday that they sign in at their designated place.

#### WHAT IF YOU HAVE QUESTIONS, SUGGESTIONS, CONCERNS, OR COMPLAINTS?

Before you decide whether to accept this invitation to take part in the study, please ask any questions that might come to mind now. Later, if you have questions, suggestions, concerns, or complaints about the study, you can contact the investigator, Dawn Brewer, PhD, RDN, LD at 859-257-1661. If you have any questions about your rights as a volunteer in this research, contact the staff in the Office of Research Integrity between the business hours of 8am and 5pm EST, Mon-Fri at the University of Kentucky at 859-257-9428 or toll free at 1-866-400-9428. We will give you a signed copy of this consent form to take with you.

# WHAT IF NEW INFORMATION IS LEARNED DURING THE STUDY THAT MIGHT AFFECT YOUR DECISION TO PARTICIPATE?

If the researcher learns of new information in regards to this study, and it might change your willingness to stay in this study, the information will be provided to you. You may be asked to sign a new informed consent form if the information is provided to you after you have joined the study.

# POTENTIAL FUTURE USE

# **Contacting Research Subjects for Future Studies**

| Do you give your permission to be contacted in the future by Dawn Brewer regarding your willingness to participate in future research studies about how to prevent, detect, or treat chronic diseases? | | | | | | |
|---|---|---|---|---|---|---|
| | Yes | | No | | _Initials | |
| Do you give your permission for photographs of you to be used on social media for promoting and advertising this program to the community? | | | | | | |
| | Yes | | No | | _Initials | Si . |
| Do you give your permission for the walking group leader to keep your contact information on file in case she needs to contact you about walking group changes, cancellations, or other updates? | | | | | | |
| | Yes | | No | | _Initials | |
| IF YES: | | | | | | |
| Na | me: | | | | g | |
| Address: | | | | | | |
| E-mail Address: | | | | | | |
| Phone Number; | | | | | | |
| WHAT ELSE DO YOU NEED TO KNOW? | | | | | | |
| There is a possibility that the data collected from you may be shared with other investigators in the future. If that is the case the data will not contain information that can identify you unless you give your consent/authorization or the UK Institutional Review Board (IRB) approves the research. The IRB is a committee that reviews ethical issues, according to federal, state and local regulations on research with human subjects, to make sure the study complies with these before approval of a research study is issued. | | | | | | |
| The National Institute of Health (NIH) is providing financial support and/or material for this study. | | | | | | |
| Signature of person agreeing to take part in the study Date | | | | | | |
| Printed name of person agreeing to take part in the study | | | | | | |
| Na | me of [autho | rize | d] person ob | taining info | rmed consent | Date |
| Signature of Principal Investigator or Sub/Co-Investigator | | | | | | |

1. **Background:** The Tanglewood Trail walking group is a community-initiated walking group, spontaneously established in summer 2016. Community members meet at the Housing Authority in Whitesburg, KY and walk the approximately 1 kilometer Tanglewood Trail connecting the Housing Authority to the Farmer's Market. Participation in the walking group is open to the public. Participants that walk to the Farmer's Market on Wednesday evenings receive a \$5 voucher to the Farmer's Market and a \$10 voucher on Saturdays during the season (June-October). Adults 18 years and older receive one voucher each time they walk. Currently, there is no evaluation of the walking group program beyond the community tracking the name, number of walkers, and the number of vouchers distributed to walkers on each Wednesday and Saturday. This program was initiated by community members and UK researchers were not involved with its creation or tracking any component of the program.

The current proposed study will target non-pregnant healthy, 18+ years old, community members who are willing and able to walk the Tanglewood Trail on Saturday mornings, June-August 2017. Community members will be randomized into a walking group and a farmers market group. Both groups will receive farmers market vouchers of equivalent value. One group will meet at the Housing Authority and walk to the farmers market to obtain their vouchers and the other group will obtain their farmers market voucher at the farmers market. Both groups are welcome to walk the Tanglewood Trail if they would like, however those that are randomized into the walking group are expected to walk. However, people are not forced to walk and have the option to refuse to walk. We hypothesize that adults who regularly attend the walking group and subsequently purchase fruits and vegetables at the Farmer's Market will experience an increase in physical activity, fruit and vegetable intake, and community engagement, and a decrease in anthropometrics and biomarkers associated with adulthood chronic disease (including cholesterol, hemoglobin A1c, blood pressure, carotenoid status, weight, and waist circumference) beyond that of the farmers market voucher group only.

# 2. Objectives:

- a) To educate Tanglewood Trail program participants about the health benefits of consuming a variety of fruits and vegetables, being physically active, and dietary strategies that can help protect their health from environmental pollution.
- b) Assess self-reported behavior change, knowledge change, and change in physical measurements (see below), and level of physical activity.
- 3. **Study Design:** The sample population consists of a convenience sample that is participating in a prospective study. This study will focus on nonpregnant healthy adult (ages 18+) community members who walk the Tanglewood Trail on Saturdays, June-August 2017.
  - Any interested community members who are 18 years or older, nonpregnant and able to voluntarily give their consent are welcome to join the study. One hundred participants will be randomized into one of two groups a walking group and a farmer's market group.
  - The fifty participants randomized into the walking group will meet at the Housing Authority at a designated time each Saturday. When they arrive, they will be signed in by a community leader and receive a farmer's market voucher (see attached) for \$10 along with education material (5 of the 13 Saturdays). They will walk as a group to the farmer's market and hand their voucher to the market manager, who will give them \$10 in tokens to purchase fruits and vegetables at the market. The voucher will have two sides: one side will ask participants what fruits and vegetables they ate the past week; the second side will ask participants to check off what fruits and vegetables they purchase at the market that day. They will turn this in as they leave the market. The fifty participants randomized into the farmer's market group will meet at- the farmer's market and sign in with a UK employee. They will receive the same voucher and education materials and follow the same procedure as the walking group. Participants randomized into this group will be allowed to walk if they want; no one will be dissuaded from engaging in physical activity. However, in order to receive their voucher, it is not required for them to walk.

Three times per month participants will be presented with education material concerning phytonutrients, the importance of fruit and vegetable intake, and how these factors might protect them from environmental pollutants. The education materials will be in the form of a.) a handout based on the Transtheoretical Model

(see attached example) or b.) Plate it Up Kentucky Proud recipe samples and cards (see attached example). A Registered Dietitian will be available to answer nutrition-based health questions once per month.

No participants will receive medications – neither real nor placebo.

Data will be a time series collection of finger-stick total cholesterol, LDL, HDL, triglycerides, hemoglobin A1c (cardiocheck meter), height, weight, waist circumference, carotenoid status (carotenoid RS, which is a non-invasive instrument that is a reliable indicator of fruit and vegetable intake (see attached), and a survey (see attached). Measurements will be taken twice – baseline data will be collected in May 2017, with follow-up data collected in early September 2017.

Finger stick tests will be conducted by University of Kentucky employees who have completed all necessary biohazard training (see attached IBC approval and certificates of completion). Lysol wipes will be available to wipe down equipment as needed. Hand sanitizer will be provided to each researcher to use between glove changes. Gloves will be changed between each participant. Heat packets will be available for participants with cold hands to make the finger stick go faster and easier. Lancets will be used to take the finger stick and all materials will be disposed of in sharps containers. All sharps containers will remain sealed until the research team returns to the University of Kentucky that same day to dispose of the sharps containers.

- 4. **Study Population:** Based on walking group numbers from summer 2016 we anticipate a maximum enrollment of 100 participants (18+ years old, nonpregnant). Previous research in Letcher County suggests the majority of participants will be white, ages 18-65, both male and female, of moderate health status. A prerequisite for participating in this study is the ability to walk approximately 1 kilometer to the Farmer's Market, nonpregnant, pre-supposing a baseline health status. Any interested community members over the age of 18 and in moderate or good health will be included. Since our focus is on changes in rates of chronic disease in adulthood, children will be excluded from study participation (but may walk the trail with their parents). Institutionalized adults, pregnant adults adults with impaired consent capacity, and prisoners will be excluded. No one will be excluded based on sex/gender or racial/ethnic identity.
- 5. Subject Recruitment Methods and Privacy: A community leader will build a facebook group in April 2017 to help recruit subjects. Interested participants will be invited to an opening baseline data collection event in May 2017. Interested participants will be told about the study and that their involvement is completely voluntary. We will obtain consent from those that are interested in participating in the study. We will then invite consented participants to fill out a survey and have the above measurements (see section 3) taken in return for a farmer's market t-shirt. Participants will be randomized into one of the two groups, walking group or farmers market only group, and informed of their group in May, during baseline measurements.

Privacy will be maintained through de-identification of all survey and measurement data. The surveys and measurement data sheets will contain a cover sheet that has a place to record the participant's name. The next page will be where the first question is listed and a space for the survey code to be recorded. Once the survey has been coded the cover sheet will be removed from the post-surveys and shredded. Participants will be asked to indicate which fruits and vegetables they purchased at the market on shopping card (**see attached**). The card will have a place for their name and they will give them to the community leader before leaving the market. The community leader will collect these weekly and give them to UK researcher bi-weekly. The shopping card data will be matched to participants' measurement data on an electronic datasheet. Once all of the data has been collected in September the electronic list of names will be replaced with a code to de-identify participants, the cover sheets of the surveys that contain participant names will be shredded and the surveys and shopping cards will be stored securely in a locked drawer in the PI's locked office. The electronic data that is generated will be stored on a password protected computer. Throughout the study, any study materials that contain participant names will be stored in a locked filing cabinet in the PI's locked office. In the event this data is published it will be done so by aggregating the data without identifying individuals.

6. **Informed Consent Process**: All study personnel that will obtain consent are listed in Form A. Participants will be told they can decide to stop their participation at any time. The consent form will be read to any study participants with visual issues. UK study personnel will speak to study participants at an appropriate volume to be heard by study participants. Study personnel will ask if they are speaking loud enough, they will tell study participants to let them know when they need to speak up or slow down or repeat a question, and study personnel will be in tune to signs of study participants straining to hear.

Consent will be obtained before physical measurements or survey data is collected. To obtain consent the UK study personnel will ask potential participants if they would like to participate in a research study that involves asking them questions about their health and diet and will also involve education material on phytonutrients, the importance of fruits and vegetables, and how these factors might protect them from environmental pollution. They will be told their participation is completely voluntary, and that they will be randomized into one of two groups. They will be informed that even if they are randomized into the farmer's market group, they are still allowed to walk whenever and however often they like. Those randomized to the walking group will be told that they are expected to walk each Saturday morning, but they will never be forced to walk and will be encouraged to abstain from walking on Saturdays when they do not feel well. They will also be told their survey answers will not be reported individually or with their name, but as anonymous aggregated data. Additionally, they will be told their participation is voluntary and they can withdraw from the study at any time and they do not have to answer any questions that they are not comfortable answering. If the participant agrees the consent form will be given to them and their signature obtained. The participant will be given a copy of an investigator-signed consent form.

The UK study personnel will ask if the participant would like to move elsewhere to complete the survey and anthropometric/biological data collection. Study personnel will also explain that the consent forms and surveys will be stored separately in a locked drawer in the PI's locked office and that an electronic file will be created that lists their name and survey code. This list will be destroyed following the collection and entry of post-survey data. Any electronic files generated from this study will be stored on a password protected computer.

Obtaining consent and completing the survey will take approximately 15 minutes. An additional 30 minutes will be needed to complete the anthropometric and biological measurements.

The midline and post data will be collected in the same manner as the pre data. The UK study personnel will offer the same explanation of the survey and anthropometric/biological measurements and the same procedures will be followed, consent however will not be obtained again. The midline and post-surveys will contain a cover sheet that has a place to record the participant's name. The next page will be where the first question is listed and a space for the survey code to be recorded. Once the survey has been coded the cover sheet will be removed from the midline and post-surveys and shredded once all data has been entered electronically.

7. Research Procedures: Following IRB approval, beginning in May 2017 community members will show up to a designated location approximately 1 kilometer from the Farmer's Market. Participants will fill out a survey and have anthropometric and biological measurements taken. Carotenoid status will be measured via carotenoid RS scanner. Anthropometric data will be collected by UK researchers and include weight (digital scale), height (portable stadiometer), waist circumference (tape) and blood pressure (digital blood pressure machine) Finger stick tests will be conducted by University of Kentucky employees who have completed all necessary biohazard training. Lysol wipes will be available to wipe down equipment as needed. Hand sanitizer will be provided to each researcher to use between glove changes. Gloves will be changed between each participant. Heat packets will be available for participants with cold hands to make the finger stick go faster and easier. Lancets will be used to take the finger stick and all materials will be disposed of in sharps containers. All sharps containers will remain sealed until the research team returns to the University of Kentucky that same day to dispose of the sharps containers.

In June through August 2017, participants in the walking group will continue to show up to the same location, be signed in by a community member, and walk approximately 1 kilometer to the Farmer's Market, in exchange for \$10 they can spend at the market. Participants in the farmer's market group will show up to the farmer's market, be signed in by a UK employee, and follow the same voucher protocol as the walking group. Three Saturdays of each month, participants from both groups will receive education material in the form of a.) handouts based on the Transtheoretical Model or b.) Plate it Up Kentucky Proud recipes samples and cards. A Registered Dietitian Nutritionist will be available at least one weekend of each month to answer nutrition-related questions.

Post-data will be collected in September 2017; the same survey will be administered and participants will again have their anthropometric and biological measurements taken.

No clinical care will be given as a part of this research study.

#### 8. Resources:

PI – Dawn Brewer, PhD, RDN, LD Program Manager – Annie Koempel, RDN, LD Research assistant – Kelci McHugh Undergraduate research assistants Community Leader Community Stakeholder

The PI, program manager, and research assistant will be responsible for all data collection and analysis. All education materials will be developed by the program manager and research assistant with oversite by the PI. The program manager and undergraduate research assistants will be USDA Good Agricultural Practices (GAP) trained to serve Plate it Up Kentucky Proud samples at one Farmer's Market per month. Undergraduate research assistants will also assist in data entry as needed (they will complete CITI certification and be added to research personnel list before having access to data). The PI will provide guidance through the process. The PI has space to store all of the consent forms, paper surveys, shopping cards and measurement data sheets in a locked drawer in the PI's locked office. All UK study personnel have computers and statistical analysis software to carry out research procedures, which are all password protected to secure any electronic files that are generated from this study. The PI has funds to purchase paper and food supplies and transportation to conduct the study.

In the event that unanticipated problems or noncompliance issues occur or the situation arises that requires submission of protocol modifications or interim results, the PI will first consult the Office of Research Integrity's website to determine action steps appropriate to the issue. If the PI still has questions she will contact the Office of Research Integrity to obtain the appropriate protocol to resolve a situation.

#### 9. Potential Risks:

No physical, psychological, social, legal, cultural, or financial risks can be perceived from participating in this research. In the rare case that a dangerously high blood pressure or hemoglobin A1c is recorded, the participant will be referred immediately to the local emergency department for care. All foods prepared for the farmer's market will be accompanied by a recipe card with ingredients. Potential allergens will be identified and communicated to all participants. Participants will not be forced to taste any food. Undergraduate research assistants will be GAP trained and knowledgeable about food safety issues. No participants will be discouraged from walking to the farmer's market, regardless of which group they are randomized into. The only difference between the two groups is where they sign in; the walking group signs in 1 kilometer from the market, while the farmer's market group signs in at the market.

Finger stick tests will be conducted by University of Kentucky employees who have completed all necessary biohazard training. Lysol wipes will be available to wipe down equipment as needed. Hand sanitizer will be provided to each researcher to use between glove changes. Gloves will be changed between each participant. Heat packets will be available for participants with cold hands to make the finger stick go faster and easier. Lancets will be used to take the finger stick and all materials will be disposed of in sharps containers. All sharps containers will remain sealed until the research team returns to the University of Kentucky that same day to dispose of the sharps containers.

A potential risk is a breach of confidentiality, which is minimal due to the study being voluntary, removing the signed consent form from the coded survey, shredding the cover sheet that contains names on the post-surveys, storing shopping cards in a locked drawer in the PI's locked office, deleting the document containing participant names and codes once the post-survey data has been coded, using a password protected computer, and storing any hard copies of study-related material in a locked drawer that is in a locked office.

10. **Safety Precautions:** Participation in every aspect of the intervention is voluntary. Participants do not have to respond to any survey questions that they are uncomfortable answering or participate in any anthropometric or biological measurements they are uncomfortable with. No one will be discouraged from engaging in physical activity.

When identifiable data (names) is being collected it will be on the cover sheet or consent form of a survey and will be detached from survey data that will include a code that is linked to the participant. At the end of the study, the cover sheets will be deleted and consent forms will be stored separately from the surveys in a locked drawer in the PI's locked office. The electronic list containing the names and survey codes will be deleted once all post-survey data is entered, which will be entered within a month following collection. However, the assigning of codes, and generating the electronic document that lists codes and names from surveys will occur the day of data collection at UK.

The study population consists of adults ages 18 years or older who are in good enough health to walk 1 kilometer to the farmer's market.

Finger stick tests will be conducted by University of Kentucky employees who have completed all necessary biohazard training. Lysol wipes will be available to wipe down equipment as needed. Hand sanitizer will be provided to each researcher to use between glove changes. Gloves will be changed between each participant. Heat packets will be available for participants with cold hands to make the finger stick go faster and easier. Lancets will be used to take the finger stick and all materials will be disposed of in sharps containers. All sharps containers will remain sealed until the research team returns to the University of Kentucky that same day to dispose of the sharps containers.

11. **Benefit vs. Risk:** Potential benefits include (but are not limited to) a decreased risk for high blood pressure, high blood glucose, and cardiovascular disease; a decrease in oxidative stress; a decrease in generalized inflammation; an increase in community engagement; an increase in physical activity, and an increase in overall fruit and vegetable consumption.

There is no more than minimal risk to participants in this intervention with the benefits outweighing any risk. There is however, a potential risk of a breach in confidentiality, which is minimal due to the study being voluntary, removing the signed consent form/cover sheet from the coded pre/post surveys, deleting the document containing participant names and codes once the post-survey data has been coded, shredding the cover sheets attached to post-surveys with participants names, using a password protected computer, and storing any hard copies of study-related material in a locked drawer that is in a locked office.

12. Available Alternative Treatment(s): N/A

13. **Research Materials, Records, and Privacy:** Participants will be asked to fill out two surveys (May and September 2017). The surveys contain questions about demographics, self-reported health, physical activity, fruit and vegetable consumption, and community engagement.

Participants will be asked to complete weekly shopping cards that will require them to mark which fruits and vegetables they purchased at the farmer's market and what fruits and vegetables they are over the past week.

Participants will be asked for finger-stick total cholesterol, LDL, HDL, triglycerides, hemoglobin A1c (cardio check meter), height, weight, waist circumference, and carotenoid status (carotenoid RS, which is a non-invasive instrument that is a reliable indicator of fruit and vegetable intake) twice (May and September 2017).

The collected data will be collated and summarized without identification or attribution to the individual participants. All reports will only reveal aggregated summaries across participants. The surveys with attached consent forms will be collected and stored separately in a locked drawer in the PI's locked office. An electronic document containing participant name and code will be generated and stored on a password protected computer. Following the collection of post-survey data and coding of the post-survey data the electronic document containing the names and codes will be deleted. To minimize risk of identification the consent forms will be removed from the survey and the survey will have a code written on it. The consent forms, shopping cards and surveys will not be stored together, but both will be in a locked drawer.

The information collected will be used to assess whether walking 1 kilometer to the farmer's market and spending approximately \$10 at the market improves physical activity, fruit and vegetable intake, community engagement, and chronic disease-related biomarkers (i.e. cholesterol, A1c, etc).

- 14. **Confidentiality:** The collated data will only reveal summarized data without identifiable information. The de-identified data will be available electronically and stored on a password protected computer. The electronic document containing names with respective survey codes will be deleted after post-survey data has been collected and therefore will not be stored. The list will be deleted by January 2020. Any study materials and raw data will be retained for 6 years in a locked drawer within a locked office or on a password protected computer. The PI and program manager assigned to the project and involved in data collection will have access to these items.
- 15. **Payment**: Participants will be offered a farmer's market t-shirt at the baseline data collection time (May 2017) and a \$10 gift card at post-data collection (September 2017) as well as the weekly \$10 voucher to the farmer's market.
- 16. Costs to Subjects: N/A
- 17. **Data and Safety Monitoring:** N/A the study does not have greater than minimal risk.
- 18. **Subject Complaints:** Participants can voice their concerns to the PI, Co-PIs, program manager, or the Office of Research Integrity, which is listed on the consent form.
- 19. Research Involving Non-English Speaking Subjects or Subjects from a Foreign Culture: N/A
- 20. HIV/AIDS Research: N/A
- 21. PI-Sponsored FDA-Regulated Research: N/A

# Tanglewood Trail Walking Program in Rural Kentucky 2017 - SAP

Analyses were conducted using SAS v. 9.4 software. For the purposes of analyses, participants were categorized as low-engagers and high-engagers defined by a cut-point of having walked to the market three or more times during the program. High-engagers were those that walked 9.0±17.2 times to the market and redeemed their vouchers 13.0±14.4 times throughout the 16-week study (n= 60). Low-engagers were those that walked 1.0±0.47 times to the farmers market and redeemed their vouchers 11.0±37.0 times (n=61).

Means and standard deviations or frequencies were calculated for each of the variables and measurements. Pre- to post-intervention differences within each group were examined using dependent t-tests and chi-square analyses as appropriate.

Repeated measures ANOVA were conducted to compare the changes in measurements including over time. Outcome variables included the finger-stick measurements, WC, BMI and blood pressure. Because fruit and vegetable consumption and physical activity are associated with improving blood lipids, blood pressure, glucose control and weight were included as independent variables in repeated measure analyses to determine if the significant changes in physical measurements were associated with fruit and vegetable consumption, walking or both. For each outcome variable, the following independent variables were included separately resulting in three different ANOVA-repeated measures analyses for each outcome variable: 1) the difference in self-reported fruit and vegetable intake from pre- to post-intervention; 2) voucher redemption rate; and 3) walking status (walked to the market  $\geq$ 3 times or <3 times throughout duration of program). If any significant associations were detected then age, sex and race were added to analyses as independent variables. Significance level was set *a priori* at p <0.05 for all analyses.